CLINICAL TRIAL: NCT04564638
Title: Long-term Outcome of Patients With Acute Ulcerative Colitis After First Course of Intravenous Corticosteroids
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Heli T Eronen, MD, specialist in internal medicine and gastroenterology, Tampere University Hospital
Other Study IDs: R15518S
Record Dates: First submitted 2020-09-11; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Ulcerative Colitis
Keywords: corticosteroids, cyclosporine, colectomy, clinical outcome
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adrenal Cortex Hormones; Cyclosporine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Corticosteroid
  Other Names: cyclosporine

SUMMARY:
All episodes of patients with acute UC admitted to Tampere University Hospital and treated with intravenous corticosteroids between January 2007 and January 2016 were identified from patient records and reviewed. The risks for colectomy and for continuous use of corticosteroids were evaluated. Predictive factors were analysed.

DETAILED DESCRIPTION:
Data collected included epidemiological (gender, age at index flare, smoking status), clinical (UC duration, extent of the disease, prior Cs usage, disease severity, laboratory results at index flare) and treatment data (occurrence of new flares, need for further Cs therapy; CyA, thiopurines, biologics or colectomy during follow-up). The diagnosis of UC was made on basis of clinical history, symptoms, endoscopic and histological features. Disease extent was categorized by the Montreal classification and the severity of the flare was assessed by Mayo scoring system based on clinical and endoscopic characteristics. ASUC was characterized by more than six bloody stools/day along with any of the following: tachycardia, elevated temperature, anemia and/or ESR >30 mm/h (Truelove and Witt´s criteria)5. Alleviation of UC was defined as clinical response to intravenous corticosteroids with no need for colectomy or rescue therapy at the same hospitalization as the index flare. Relapse was defined as requiring further corticosteroid treatment, rehospitalization, rescue-therapy, or colectomy later in follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Acute severe ulcerative colitis treated first time with iv corticosteroids
* Follow-up for at least six months after hospitalization or until colectomy.

Exlusion:

-Under 16 year of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients treated in hospital ward with first intravenous corticosteroid
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Colectomy | Long-term follow-up. Years 2007-2016. Mean follow-up of 7.5 years.
  We reviewed patient records for data on need for surgery within follow-up. We identified patients who had emergency colectomy and patients who needed surgery within 1 year of index flare or within follow-up.
Responce to Corticosteroid | Admission on index flare
  Responce to first intravenous corticosteroid was defined as no need for colectomy or rescue therapy within admission.

IPD SHARING:
Plan to Share IPD: Undecided